CLINICAL TRIAL: NCT03134105
Title: A Wearable EducAtional Intervention to REduce Angina
Acronym: AWARE
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsor/funding source decided to not move forward.
Sponsor: Duke University (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00081545
Record Dates: First submitted 2017-04-26; First posted 2017-04-28 (Actual); Last update posted 2017-08-21 (Actual); Status verified 2017-04

CONDITIONS: Angina
MeSH Terms: conditions — Angina Pectoris

STUDY DESIGN:
Intervention Model Description: This study will enroll patients with recent myocardial infarction being seen in cardiology clinics. All patients will receive wearable fitness trackers and apps that capture this data and transmit it to the coordinating center; patients will also provide information on angina frequency every other week via emailed surveys. Sites will be randomized to have their providers receive either monthly updates on step count and patient reported angina or a single report at the end of the study period. Providers receiving monthly reports will receive a single report with data for each of their patients participating in the study along with summary data for their practice and all patients participating in the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Monthly Feedback (Experimental): Sites will receive monthly reports of their patients enrolled in the study with data for each of their patients participating in the study along with summary data for their practice and all patients participating in the study.
  Interventions: Other: Monthly Feedback on activity and patient-reported angina
- End-of-study Feedback (Active Comparator): Sites will only receive the report of their patients at the end of the 6 month follow-up period.
  Interventions: Other: End-of-Study Feedback

INTERVENTIONS:
Other: Monthly Feedback on activity and patient-reported angina — Providers will receive monthly updates on step count and patient reported angina for each of their patients, with data derived from a wearable fitness tracker and every other week emailed surveys
  Arms: Monthly Feedback
Other: End-of-Study Feedback — Providers will receive an end-of-study update on step count and patient reported angina for each of their patients, with data derived from a wearable fitness tracker and every other week emailed surveys
  Arms: End-of-study Feedback

SUMMARY:
The AWARE-Angina study is a cluster randomized trial aimed at evaluating whether routine provider feedback of patients' angina burden and activity level can improve angina control. Patients will wear an activity monitor for 6 months, and their providers will be randomized to receive either monthly feedback or feedback at the end of the study period.

DETAILED DESCRIPTION:
This is a cluster randomized trial of using a wearable activity monitor to enhance communication between patients with recent acute Myocardial Infarction (MI) and their physicians. After IRB approval, each site will be randomly assigned to either the monthly feedback or the end-of-study feedback arm. All participating providers will participate in an accredited webinar discussing the prevalence of post-MI angina, effects of angina on quality of life and outcomes, and the evidence supporting use of available treatment options. The intention of this approach is to develop a similar baseline understanding of angina among the participants so that knowledge gaps do not interfere with the intervention described below.

Patients at each site who meet the eligibility criteria (acute MI within 6 months with documentation of at least single-vessel coronary artery disease, possession of a smartphone) will be approached for consideration of participation. Those who qualify and express interest will provide informed consent to the study procedures.

At the time of enrollment, patient data (including socio-demographic information, medial history and comorbidities, details of the patient's index MI, secondary prevention medications, and anti-anginal medication prescriptions) will be collected by participating sites for each enrolled patient via a paper data collection form and faxed to a secure fax machine at the DCRI. Patients will also complete a brief survey including questions about angina frequency and quality of life.

All patients will receive a wearable activity tracker (WithingsGO) and smartphone-based app (Withings Health mate). Patients will be instructed on how to put on and take off the wearable activity monitor. They will be instructed to wear the activity monitor continuously while awake for the duration of the study. For the next 6 months, the wearable activity monitor will measure daily step count and distance walked. This data will be transmitted continuously via a Bluetooth connection to the smartphone-based app. The activity monitor application will share activity data through Validic with DCRI IT/CDM through a secure Web Portal. Every other week, patients will receive an email with a link to a Qualtrics survey including questions regarding angina frequency, angina severity, use of short-acting nitroglycerin tablets, and whether they had any overnight hospitalizations in the 2 weeks prior. The survey data will be transmitted to the DCRI through Qualtrics. If patients miss 2 or more consecutive Qualtrics surveys, then representatives from DCRI will contact the patient to complete.

ELIGIBILITY:
Inclusion Criteria:

1. Acute MI within the prior 6 months
2. At least one-vessel coronary artery disease (≥70% obstruction in any coronary artery or ≥50% in the left main coronary artery)
3. English speaking

Exclusion Criteria:

1. Unable or unwilling to provide informed consent, including but not limited to cognitive or language barriers (reading or comprehension)
2. Non-ambulatory
3. Anticipated life expectancy less than 6 months
4. Does not own a smartphone operating the iOS or Android operating system

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-09 (Estimated); Primary Completion 2018-02 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
Change in patients' mean daily number of steps | Baseline to 6 months
  The investigator will plot step count for each patient over the study period and calculate a slope, representing change in number of steps per day enrolled in the study. The research team will calculate a mean slope for patients in each group (monthly feedback versus end-of-study period feedback) and compare between groups. 1. Number of steps will be measured continuously, and the team will evaluate the difference between baseline and 6 months

SECONDARY OUTCOMES:
Change in Distance Walked | Baseline to 6 months
  The investigator will get the daily distance walked from the start of the study to the end
Change in Angina Frequency | Baseline to 6 months
  The investigator will compare between groups the proportion of patients with a reduction in self-reported angina frequency from baseline to 6 months
Change in Anti-Anginal Medication | Baseline to 6 months
  The investigator will look at the proportion of patients initiating a new non-beta blocker anti-anginal medication from baseline to 6 months

IPD SHARING:
Plan to Share IPD: No